CLINICAL TRIAL: NCT04019028
Title: Real-time Monitoring of Motor Cortical Activity Induced by Low-frequency Repetitive Transcranial Magnetic Stimulation: Functional Near Infrared Spectroscopic Study
Brief Title: Real-time Monitoring of Motor Cortical Activity Induced by Low-frequency Repetitive Transcranial Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2014-05-021
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: low frequency rTMS; fNIRS; Hemodynamic Response; Non-invasive brain stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Navigated low frequency rTMS (Experimental): Application of 1Hz low frequency repetitive transcranial magnetic stimulation to the primary motor area of the dominant hemisphere using a navigation system.
  Using the BrainSight instrument, a navigation system, the TMS coil position can be fixed on the point precise target area based on the subject's MRI image.
  Interventions: Device: low frequency rTMS + Navigation System
- only low frequency rTMS(not using Navigation System) (Experimental): Application of low frequency repetitive transcranial magnetic stimulation to the primary motor area of the dominant hemisphere not using a navigation system.
  TMS coil is fixed on the target area based on MEP hotspot.
  Interventions: Device: only low frequency rTMS
- Navigated Sham rTMS (Sham Comparator): Application of repetitive transcranial magnetic stimulation with sham mode(no stimulation) to the primary motor area of the dominant hemisphere using a navigation system.
  Using the BrainSight instrument, a navigation system, the TMS coil position can be fixed on the point precise target area based on the subject's MRI image.
  Sham stimulation is stimulated by the same frequency, intensity and time as the actual stimulus in such a way that the 8-shaped coil is placed at a 90 degree angle to the scalp in the same manner as rTMS and sounds are heard but the magnetic stimulus is not transmitted to the cerebrum
  Interventions: Device: Sham low frequency rTMS + Navigation System

INTERVENTIONS:
Device: low frequency rTMS + Navigation System — 1Hz low-frequency rTMS stimulation over primary motor area using navigation system
  Arms: Navigated low frequency rTMS
Device: only low frequency rTMS — 1Hz low-frequency rTMS stimulation over primary motor area
  Arms: only low frequency rTMS(not using Navigation System)
Device: Sham low frequency rTMS + Navigation System — 1Hz low-frequency sham rTMS stimulation over primary motor area using navigation system
  Arms: Navigated Sham rTMS

SUMMARY:
In this study, we investigated the effect of low-frequency repetitive trans cranial magnetic stimulation, one of the noninvasive brain stimuli, on the functional changes of the bilateral motor cortical activity in normal subjects using functional near infrared spectroscopy (fNIRS).

DETAILED DESCRIPTION:
In normal subjects,

1. the effect of low-frequency repetitive transcranial magnetic stimulation on cerebral cortex are measured in real time using fNIRS.
2. Changes in cerebral cortical activity before and after stimulation are measured using the motor function test and the motor-induced potential test

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women without history of central nervous system disease and abnormalities

Exclusion Criteria:

* Under 18 years old, 70 years old or older
* A person who has inserted a metal object in a skull
* A person with complete occlusion of the carotid artery
* A person with epilepsy
* Pregnant and lactating women
* Who is not eligible for the test

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Changes of Cortical activation | Baseline and after intervention[Immediately after 20 minutes of intervention]
  Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) before and after stimulation

SECONDARY OUTCOMES:
Changes in motor evoked potentia | Baseline and after intervention[Immediately after 20 minutes of intervention]
  measure the motor threshold and amplitude of motor evoked potential in first dorsal interosseous muscle.
changes in nine hole peg test | Baseline and after intervention[Immediately after 20 minutes of intervention]
  Nine-Hole Peg Test is used to measure finger dexterity in patients with various neurological diagnoses.
Sequential motor task | Baseline and after intervention[Immediately after 20 minutes of intervention]
  It is a training exercise in which five digits are repeatedly pressed with five fingers using individual movements, and it is trained to press the button accurately and quickly.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kimm, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea